CLINICAL TRIAL: NCT03337932
Title: Duration of Doxycycline Treatment in Patients With Multiple Erythema Migrans (MEM). A Randomized Clinical Trial
Brief Title: Duration of Doxycycline Treatment in MEM Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Daša Stupica, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEM-Doxy
Record Dates: First submitted 2017-10-24; First posted 2017-11-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Erythema Chronicum Migrans
MeSH Terms: conditions — Erythema Chronicum Migrans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MEM-7 days doxycycline (Active Comparator)
  Interventions: Drug: Doxycycline 100 milligram Oral Tablet bid, 7 days
- MEM-14 days doxycycline (Active Comparator)
  Interventions: Drug: Doxycycline 100 milligram Oral Tablet bid, 14 days
- Controls (Placebo Comparator)
  Interventions: Drug: Controls without a history of lyme disease.

INTERVENTIONS:
Drug: Doxycycline 100 milligram Oral Tablet bid, 7 days — Patients will receive doxycycline for 7 days.
  Arms: MEM-7 days doxycycline
Drug: Doxycycline 100 milligram Oral Tablet bid, 14 days — Patients will receive doxycycline for 14 days.
  Arms: MEM-14 days doxycycline
Drug: Controls without a history of lyme disease. — No intervention.
  Arms: Controls

SUMMARY:
The purpose of this study is to compare the efficacy of 7-day versus 14-day doxycycline treatment in patients with multiple erythema migrans.

ELIGIBILITY:
Inclusion Criteria:

• multiple erythema migrans

Exclusion Criteria:

* pregnancy or lactation
* immunocompromised
* serious adverse event to doxycycline
* taking antibiotic with antiborrelial activity within 10 days
* extracutaneous manifestations of lyme borreliosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 14 days post-enrollment in patients treated for multiple erythema migrans with doxycycline for 7 or 14 days | Study point: at 14 days post-enrollment.
  At follow-up at 14 days patients will be examined physically and will be asked an open question about health-related symptoms. Symptoms that will newly develop or worsen since the onset of the multiple erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis will be interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 2 months post-enrollment in patients treated for multiple erythema migrans with doxycycline for 7 or 14 days | Study point: at 2 months post-enrollment.
  At follow-up at 2 months patients will be examined physically and will be asked an open question about health-related symptoms. Symptoms that will newly develop or worsen since the onset of the multiple erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment will be interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 6 months post-enrollment in patients treated for multiple erythema migrans with doxycycline for 7 or 14 days | Study point: at 6 months post-enrollment.
  At follow-up at 6 months patients will be examined physically and will be asked an open question about health-related symptoms. Symptoms that will newly develop or worsen since the onset of the multiple erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment will be interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 12 months post-enrollment in patients treated for multiple erythema migrans with doxycycline for 7 or 14 days | Study point: at 12 months post-enrollment.
  At 12 months patients will be examined physically and will be asked an open question about health-related symptoms. Symptoms that will newly develop or worsen since the onset of the multiple erythema migrans and which will have no other known medical explanation will be regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment will be interpreted as failure.

SECONDARY OUTCOMES:
Change in occurrence of nonspecific symptoms from baseline to 6 months and to 12 months post-enrollment in patients with multiple erythema migrans and control subjects | Study points will be: at enrollment, at 6, and at 12 months post-enrollment.
  Patients will complete a written questionnaire asking whether they had had any of 8 nonspecific symptoms (fatigue, arthralgias, headache, myalgias, paresthesias, memory difficulties, concentration difficulties, irritability) within the preceding week.
  Control subjects will complete the same 8-symptom questionnaire as the patients within 14 days of the examination date of the corresponding patient at enrollment, and again at 6 and 12 months.
  Patients and controls will grade the severity of each individual symptom on a 10-cm visual analogue scale (10 = most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Daša Stupica, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical center Ljubljana, Ljubljana, Slovenia